CLINICAL TRIAL: NCT03332251
Title: Anisotropic Textile Braces for Adolescent Idiopathic Scoliosis
Brief Title: Trial of Posture Correction Girdle for Adolescents With Early Scoliosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Joanne Yip, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GRF2017
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Scoliosis
Keywords: Posture Correction Girdle
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Posture Correction Girdle (Experimental): The design of posture correction girdle will incorporate different mechanisms, such as a) compression and pulling forces through a close fit of the intimate apparel, b) lumbar flexion by using a supporting belt, c) transverse forces applied by inserting pads inside the pocket lining by using the principle of the 3-point pressure system, d) axial rotation or coupled motion by using a system with uneven straps, and e) an active mechanism that aims to shift the trunk away from areas of pressure
  Interventions: Device: Posture Correction Girdle
- Control (No Intervention): No treatment will be provided for control participants.

INTERVENTIONS:
Device: Posture Correction Girdle — Participants will be invited to undergo a fitting session of posture correction girdle. After the fitting, participants will join a 6-month wear trial of the posture correction girdle. Participants are required to wear the girdle for 8 hours a day and the compliance will be recorded by a logbook daily. Participants will be invited to undergo assessments before the wear trial, after the trial of 3 months, and after the trial of 6 months. The measure outcomes of the assessment include 1) ultrasound scanning image, 2) 3D body scan, 3) electromyography signal, 4) garment pressure, and 5) questionnaire.
  Arms: Posture Correction Girdle

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a prevalent chronic condition that gradually leads to the three dimensional deformity of the spine. Spine curvature increases in youths as puberty progresses. Generally, only observation is suggested for adolescents with early scoliosis (Cobb's angle ≤ 20°). Rigid brace treatment is too draconian for them due to the high corrective force which nearly constrains all movements. Flexible brace treatment is an alternative option; however, its efficacy is still controversial. Posture correction girdle with a specialized design for teenagers with scoliosis is limited and most part of them can only provide some improvement for bad postures, such as hunchback. A scientific approach should be used to design and develop posture correction girdle as a treatment option for adolescents with early scoliosis.

DETAILED DESCRIPTION:
The design of posture correction girdle will incorporate different mechanisms, such as

1. compression and pulling forces through a close fit of the intimate apparel
2. lumbar flexion by using a supporting belt
3. transverse forces applied by inserting pads inside the pocket lining by using the principle of the 3-point pressure system
4. axial rotation or coupled motion by using a system with uneven straps, and
5. an active mechanism that aims to shift the trunk away from areas of pressure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS
* Cobb's angle 10˚-20˚
* Risser grade ≤ 2
* No prior treatment
* Pre-menarche or post- menarche by no more than 1 year
* Ability to read and understand English or Chinese
* Physical and mental ability to adhere to anisotropic textile braces protocol

Exclusion Criteria:

* Diagnosis of other musculoskeletal or developmental illness that might be responsible for the spinal curvature
* History of previous surgical or orthotic treatment for AIS
* Contraindications for pulmonary and/ or exercise tests
* Psychiatric disorders
* Recent trauma
* Recent traumatic (emotional) event

Ages: 10 Years to 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of posture correction girdle | 6 months
  The spinal curve progression is said to be under control if the increase in the Cobb's angle is <5°

SECONDARY OUTCOMES:
Posture improvement | 6 months
  Improvement of posture by clinical photographs assessment

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China